CLINICAL TRIAL: NCT04335526
Title: A Clinical Study for Assessing the Effect of Change of Bile Acid Pool on the Pharmacodynamics and Safety of Metformin and Intestinal Microbiome Profiles in Healthy Volunteers
Brief Title: A Clinical Study to Assess the Effect of Change of Bile Acid on the PD and Safety of Metformin and Microbiome Profiles
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae Yong Chung, MD, PhD, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MMP2
Record Dates: First submitted 2020-04-03; First posted 2020-04-06 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Human Microbiome
MeSH Terms: interventions — Cholestyramine Resin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin alone (No Intervention)
- Metformin with cholestyramine (Other)
  Interventions: Drug: Cholestyramine Resin

INTERVENTIONS:
Drug: Cholestyramine Resin — Change bile acid pool by cholestyramine treatment
  Arms: Metformin with cholestyramine

SUMMARY:
This clinical trial is intended to evaluate the effect of change of bile acid pool with cholestyramine on the pharmacodynamics and safety of metformin and intestinal microbiome profiles in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 to 50, healthy male subjects(at screening)
* Body weight between 50.0 kg - 100.0 kg, BMI between 18.0 - 28.0 kg/m2
* Subject who totally understand the progress of this clinical trials, make decision by his free will, and signed a consent form to follow the progress

Exclusion Criteria:

* Subject who has a past or present history of any diseases following below.(liver, kidney, neurology, immunology, pulmonary, endocrine, hematology, oncology, cardiology, mental disorder)
* Subject who had GI tract disease(Crohn's disease, ulcer, acute or chronic pancreatitis) or surgery (appendectomy, hernioplasty are excluded)
* Serum AST(SGOT), ALT(SGPT)>2 times upper limit of normal range MDRD eGFR <80mL/min/1.73m2
* Subject who had drug (Aspirin, antibiotics) hypersensitivity reaction
* Subject who already participated in other trials in 3 months
* Subject who had whole blood donation in 2 months, or component blood donation in 1 month or transfusion in 1 month currently

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Compare the maximum blood glucose concentration (Gmax) | Day 1/2/8/9 (pre-dose (75 g glucose), 0.25, 0.5, 0.75, 1, 1.5. 2 hours)
  Compare the maximum blood glucose concentration (Gmax) between meformin alone and meformin with cholestyramine
Compare the maximum blood glucose concentration (Gmax) | Day 1/2/8/9 (pre-dose (75 g glucose), 0.25, 0.5, 0.75, 1, 1.5. 2 hours)
  Compare the area under the blood glucose concentration versus time curve (AUC) between meformin alone and meformin with cholestyramine
Compare the gut microbiome species change | Day 1/2/8/9
  Compare how the gut microbiome species change between meformin alone and meformin with cholestyramine

CONTACTS AND LOCATIONS:
Overall Officials: Chung Jae Yong, MD, PhD, Principal Investigator — Department of Clinical Pharmacology and Therapeutics, Seoul National University College of Medicine and Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided